CLINICAL TRIAL: NCT05253352
Title: Variable Anatomy and Function of the Arm's Alternate Lymphatic Pathway
Brief Title: Mapping and Quantifying Lymphatic Drainage of the Arm's Alternate Pathway
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dhruv Singhal, Associate Professor, Beth Israel Deaconess Medical Center
Other Study IDs: 2021P000209; 1R01HL157991-01 (NIH)
Record Dates: First submitted 2022-02-11; First posted 2022-02-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Lymphatic System
Keywords: anatomy; lymphatic system

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy volunteers: Healthy female volunteers with no history of lymphedema. Physical therapy examination, ICG lymphography, venous ultrasound and lymphoscintigraphy with SPECT/CT imaging
- Women with breast cancer who did not develop lymphedema: Women who have had an axillary lymph node dissection (ALND) and did not develop lymphedema. Physical therapy examination, ICG lymphography, venous ultrasound and lymphoscintigraphy with SPECT/CT imaging

SUMMARY:
Using indocyanine green (ICG) lymphography and lymphoscintigraphy with SPECT/CT imaging, the aim is to evaluate the anatomy of the lymphatic system pathway in two separate populations: healthy female volunteers and women with a history of breast cancer who did not develop lymphedema.

DETAILED DESCRIPTION:
Breast Cancer Related Lymphedema (BCRL) affects 1.2 million patients in the United States and has no cure. The symptoms of lymphedema include fatigue, tightness, pain, and life-threatening infections. However, two-thirds of women undergoing breast cancer treatment with the highest risk factors for developing lymphedema do not develop the disease. While there is no explanation for this finding, one hypothesis is that normal anatomic variations of the lymphatic system pre-dispose certain women to developing lymphedema after breast cancer treatment. Specifically, the main back-up lymphatic pathway of the arm, the Mascagni-Sappey (M-S) pathway, is variably present in cadaver studies and avoids areas that are usually damaged with breast cancer treatment. Moreover, when present in these cadaver studies, the M-S pathway has variable anatomic connections which can impact its ability to drain the arm effectively. The investigators hypothesize that, utilizing modern imaging techniques, the investigators can define the anatomy of the M-S pathway and its variations in normal women and in breast cancer survivors who have undergone high risk breast cancer treatment and did not develop lymphedema. Utilizing this information, the investigators will be able to predict which variations predispose women to develop lymphedema. Finally, the investigators will develop a novel method of non-invasive intraoperative optical imaging to assess the function of this pathway during breast cancer operations to predict the patient's risk of developing lymphedema. The ability to evaluate real-time lymphatic function would allow cancer teams to implement preventive interventions in high risk patients. As the most common cause of lymphedema in the United States is secondary to cancer procedures, this model of lymphedema prevention could be widely applied to the treatment of other high risk cancer populations including gynecologic cancers, urologic cancers, skin cancers, and sarcomas.

The investigators will use ICG lymphography and lymphoscintigraphy with SPECT/CT (single-photon emission computed tomography) imaging to evaluate the anatomy of the M-S pathway in two separate populations:

Group 1: The research study staff will recruit healthy female volunteers without a history of lymphedema or ALND (axillary lymph node dissection) surgery to map the normal anatomy of the M-S pathway. The investigators hope to quantify the percentage of women who do not have this pathway present, do not have peripheral connections between the M-S pathway and the forearm, and/or whose terminal M-S pathway draining nodal basins are in the axilla.

Group 2: Research study staff will measure changes that occur in the M-S pathway anatomy in women at least 2 years status-post ALND surgery without developing lymphedema in the time following their surgery (Aim 2) using the same methodology. By understanding the M-S pathway anatomy in relation to the main lymphatic drainage pathway of the forearm in the setting of an ALND without lymphedema the investigators can gain critical insight about which patients are at the highest risk of developing BCRL and why this is more likely to occur in some patients than others.

ELIGIBILITY:
Inclusion Criteria:

* Female
* History of breast cancer treatment including ALND - defined by removal of >=10 lymph nodes - more than 2 years before study participation
* Ability to understand the protocol and willingness to participate
* At least 18 years of age

Exclusion Criteria:

* Prior history of bilateral lymph node surgery
* Prior history of other surgical procedures of the affected upper extremity besides the axillary management for breast cancer treatment
* Prior history of chronic inflammatory conditions (e.g. rheumatoid arthritis)
* Prior history of filarial infections
* Prior history of lymphedema
* Patient-reported pregnancy
* Patients who are breastfeeding
* Iodine allergy
* Prior history of upper extremity deep vein thrombosis
* Prior history of congestive heart failure
* Prior history of venous thoracic outlet syndrome
* Current active cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with a history of breast cancer treatment including axillary lymph node dissection (ALND) more than 2 years prior to study participation, who did not develop lymphedema.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lymphatic pathway anatomy of the upper extremity | Study Visit 1: Immediately after ICG lymphography injections
  Indocyanine green (ICG) lymphography of bilateral upper arms
Lymphatic pathway anatomy of the upper extremity | Study Visit 1: 30 min after lymphoscintigraphy tracer injection
  Lymphoscintigraphy scans of bilateral upper arms
Lymphatic pathway anatomy of the upper extremity | Study Visit 1: 2 hours after lymphoscintigraphy tracer injection
  Lymphoscintigraphy scans of bilateral upper arms
Lymphatic pathway anatomy of the upper extremity (SPECT/CT) | Study Visit 1: 2 hours after lymphoscintigraphy tracer injection
  SPECT/CT lymphoscintigraphy scans of bilateral upper arms
Lymphatic pathway anatomy of the upper extremity | Study Visit 2: 30 min after lymphoscintigraphy tracer injection
  Lymphoscintigraphy scans of bilateral upper arms
Lymphatic pathway anatomy of the upper extremity | Study Visit 2: 2 hours after lymphoscintigraphy tracer injection
  Lymphoscintigraphy scans of bilateral upper arms
Lymphatic pathway anatomy of the upper extremity (SPECT/CT) | Study Visit 2: 2 hours after lymphoscintigraphy tracer injection
  SPECT/CT lymphoscintigraphy scans of bilateral upper arms

CONTACTS AND LOCATIONS:
Overall Officials: Dhruv Singhal, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided